CLINICAL TRIAL: NCT02622581
Title: Clinical Research Platform Into Molecular Testing, Treatment and Outcome of (Non-)Small Cell Lung Carcinoma Patients
Acronym: CRISP
Status: Recruiting | Type: Observational
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry); Celgene Corporation (Industry); Merck Sharp & Dohme LLC (Industry); Novartis Pharmaceuticals (Industry); Pfizer (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); iOMEDICO AG (Industry); Eli Lilly and Company (Industry); Roche Pharma AG (Industry); Takeda (Industry); Amgen (Industry); Janssen-Cilag G.m.b.H (Industry); GlaxoSmithKline (Industry); Daiichi Sankyo (Industry); Regeneron Pharmaceuticals (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AIO-TRK-0315
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Non-small Cell Lung Cancer (NSCLC); Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage II; Non Small Cell Lung Cancer Stage III; Small-cell Lung Cancer; Non-small Cell Lung Cancer Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — All patients will be asked to give consent for their tumor samples to be used for future investigational translational research. If the patient agrees, contact details of the local pathology where the tumor sample is stored as well as the sample's identification number will be documented in the eCRF, creating the CRISP "decentralized clinically annotated tissue repository". Study sites will inform the local pathologists about the patient's consent and ask for the tissue sample to be reserved for future CRISP analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- NSCLC, Non-squamous cell carcinoma: Patients with locally advanced or metastatic NSCLC at the start of palliative first-line systemic therapy or receiving best supportive care.
  At least 3,250 patients with non-squamous cell carcinoma will be tested for molecular alterations. (CRISP)
  Interventions: Other: data collection
- NSCLC, Squamous cell carcinoma: Patients with locally advanced or metastatic NSCLC at the start of palliative first-line systemic therapy or receiving best supportive care.
  At least 1,750 patients with squamous cell carcinoma that possibly will be tested for molecular alterations. (CRISP)
  Interventions: Other: data collection
- NSCLC, Non-squamous cell carcinoma (not tested): Patients with locally advanced or metastatic NSCLC at the start of palliative first-line systemic therapy or receiving best supportive care.
  Up to 5,000 patients not tested for molecular alterations (CRISP satellite untested patients stage IIIB/IIIC/IV).).
  Interventions: Other: data collection
- NSCLC, Stage I/II/III: Up to 1600 patients with NSCLC stage I, or stage II, or stage IIIA, or with NSCLC stage IIIB/C if they are eligible for curative surgery and/or radiochemotherapy, or are receiving best supportive care
  Interventions: Other: data collection
- Small cell lung cancer (SCLC): Up to 1200 patients with SCLC (limited stage (LD) or extensive stage (ED)) if they are eligible for surgery and/or radio(chemo)therapy and/or systemic therapy, or are receiving best supportive care
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Baseline (demographic, clinical, tumor) characteristics, details on biomarker testing, including re-testing, treatment decision making, all systemic anticancer therapies including details, key data on radiotherapies, surgeries and specified supportive therapies, outcome (response, progression, survival), course of disease. Data will be documented at baseline and updated at least every three months.

SUMMARY:
Open, non-interventional, prospective, multi-center clinical research platform with the main objective to assess molecular biomarker testing, treatment and outcome of patients with NSCLC or SCLC in Germany

DETAILED DESCRIPTION:
Thorough knowledge of the treatment reality, e.g. characteristics, diagnostic, treatment and outcome of unselected patients in real-life practice, is crucial to evaluate and improve the quality of care for patients with non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).

The purpose of CRISP is to set up a national clinical research platform to document uniform data on the molecular testing, treatment, course of disease in patients with NSCLC or SCLC. A particular focus is on molecular biomarker testing before the start of first-line treatment of patients with advanced or metastatic NSCLC. The data shall be used to assess the current state of care and to develop recommendations concerning topics that could be improved.

PRO assessment will provide large-scale data on quality of life and anxiety/depression for real-life patients with NSCLC or SCLC in routine practice. In addition, two questionnaires (concerning individual quality of life and patient-caregiver communication) will be validated in German patients with metastatic NSCLC.

Furthermore, CRISP will set up a decentralized clinically annotated tissue repository for future collaborative, investigational scientific biomarker testing.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for the project:

* Age ≥ 18 years
* Able to understand and willing to sign written Informed Consent and to complete patient-reported-outcome assessment instruments

Main project (Metatstatic NSCLC):

* Confirmed non-small cell lung cancer (NSCLC)
* Informed consent no later than four weeks after start of first-line systemic treatment or no later than four weeks after diagnosis for patients receiving "best supportive care only"
* Stage IV, or stage IIIB/C (UICC8) if patient is ineligible for curative surgery and/or radiochemotherapy
* Systemic therapy or best supportive care

Satellite Stage I/II/III (NSCLC):

* Confirmed non-small cell lung cancer (NSCLC)
* Informed consent no later than four weeks after start of first anti-tumor treatment (including surgery and radiotherapy) or no later than four weeks after diagnosis for patients receiving "best supportive care only" (i.e. no anti-tumor treatment = no surgery, radiotherapy or systemic therapy)
* Stage I, Stage II, stage IIIA, or stage IIIB/C (UICC8)
* Systemic (chemo)therapy and/or radiation therapy and/or surgery or best supportive care

Satellite SCLC

* Confirmed Small cell lung cancer (SCLC)
* Informed consent no later than four weeks after start of first anti-tumor treatment or no later than four weeks after diagnosis for patients receiving "best supportive care only" (i.e. no anti-tumor treatment = no surgery, radiotherapy or systemic therapy)
* Systemic (chemo)therapy and/or radiation therapy and/or surgery or best supportive care

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Main project (Metastatic NSCLC):
  10000 patients with locally advanced or metastatic NSCLC at the start of palliative first-line systemic therapy or receiving best supportive care (BSC). 5000 will be patients with non-squamous cell carcinoma tested for molecular alterations at the start of first-line or patients with squamous cell carcinoma (CRISP patients). The remainder will be patients with untested non-squamous carcinoma (CRISP satellite untested patients stage IIIB/IIIC/IV).
  Satellite Stage I/II/III (NSCLC):
  1600 patients with NSCLC stage I,II,IIIA or IIIB/C eligible for curative surgery and/or radiochemotherapy or receiving BSC.
  Satellite SCLC:
  Up to 1200 patients with SCLC (limited stage or extensive stage) eligible for surgery and/or radio(chemo)therapy and/or systemic therapy or receiving BSC.
  Patients will be recruited in up to 150 study sites (certified lung cancer centers, comprehensive cancer centers, hospitals and office-based oncology practices) in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 12400 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
biomarker | 3 years
  To collect data on the frequency, methodology and results of molecular biomarker testing before first-line and later-line treatment
treatment | 3 years
  To describe systemic treatments and sequential treatments applied in real-life practice
Response rate | 3 years
  To assess effectiveness of systemic treatments in regards to response rate.
progression free survival | 3 years
  To assess effectiveness of systemic treatments in regards to progression free survival.
overall survival | 3 years
  To assess effectiveness of systemic treatments in regards overall survival.
physician-reported factors | 3 years
  To describe physician-reported factors affecting treatment decision making besides biomarker profiling
supportive therapies | 3 years
  to collect key data on specific supportive therapies
changes during the project | 3 years
  To investigate changes in diagnostics, treatment or outcome during the course of the project
general health-related and individual quality of life (QoL) patient-reported outcomes | 3 years
  To evaluate patient-reported outcomes concerning (1) general health-related and individual quality of life (QoL). and depression, (4) patient-caregiver communication
physical and psychological well-being patient-reported outcomes | 3 years
  To evaluate patient-reported outcomes concerning physical and psychological well-being.
anxiety patient-reported outcomes | 3 years
  To evaluate patient-reported outcomes concerning anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Griesinger, Prof. Dr., Principal Investigator — Pius-Hospital Oldenburg
Locations (1):
- Pius-Hospital, Oldenburg, Germany

REFERENCES:
- [Derived] Metzenmacher M, Griesinger F, Hummel HD, Elender C, Schafer H, de Wit M, Kaiser U, Kern J, Janicke M, Spring L, Zacharias S, Kaiser-Osterhues A, Groth A, Hipper A, Zaun G, Dorfel S, Guldenzoph B, Muller L, Uhlig J, Thomas M, Sebastian M, Eberhardt WEE; CRISP Registry Group. Prognostic factors in nonsmall cell lung cancer: insights from the German CRISP registry. Eur Respir J. 2023 Feb 2;61(2):2201336. doi: 10.1183/13993003.01336-2022. Print 2023 Feb. PMID 36180086
- [Derived] Griesinger F, Eberhardt W, Nusch A, Reiser M, Zahn MO, Maintz C, Bernhardt C, Losem C, Stenzinger A, Heukamp LC, Buttner R, Marschner N, Janicke M, Fleitz A, Spring L, Sahlmann J, Karatas A, Hipper A, Weichert W, Heilmann M, Sadjadian P, Gleiber W, Grah C, Waller CF, Reck M, Rittmeyer A, Christopoulos P, Sebastian M, Thomas M; CRISP Registry Group. Biomarker testing in non-small cell lung cancer in routine care: Analysis of the first 3,717 patients in the German prospective, observational, nation-wide CRISP Registry (AIO-TRK-0315). Lung Cancer. 2021 Feb;152:174-184. doi: 10.1016/j.lungcan.2020.10.012. Epub 2020 Nov 2. PMID 33358484
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — https://www.aio-portal.de